CLINICAL TRIAL: NCT04743336
Title: The Relationship Between Body Mass Index and Stage/Grade of Periodontitis
Brief Title: The Relationship Between Body Mass Index and Periodontitis
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Mehtap Bilgin Çetin, Assosc.Prof.Ph.D, Baskent University
Other Study IDs: MBÇ
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Obesity; Periodontitis
MeSH Terms: conditions — Obesity; Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal weight (<25 kg/m2)
  Interventions: Other: Measuring pocket depth
- overweight (25-29.9 kg/m2)
  Interventions: Other: Measuring pocket depth
- obese (≥30 kg/m2)
  Interventions: Other: Measuring pocket depth

INTERVENTIONS:
Other: Measuring pocket depth — Probing pocket depth (PPD = distance between gingival margin and bottom of the periodontal pocket)were evaluated in each patient. All periodontal measurements were recorded at six sites around each tooth by a periodontal probe excluding third molar

SUMMARY:
This study aimed to examine the relationship between body mass index (BMI) and stage/grade of periodontitis per the current classification of periodontal diseases.

142 patients (82 males/60 females) were included in this study. "2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions" was taken as basis to characterize the stage/grade of periodontitis. As well as age, gender, smoking status, and frequency of tooth brushing, medical data of the patients including hypertension, hyperlipidemia, BMI, and diabetes mellitus were obtained from the patient's hospital records. Obesity was assessed by BMI using the "World Health Organization" criteria.

DETAILED DESCRIPTION:
In this retrospective study, dental and medical records of 200 patients diagnosed with periodontitis who applied to Baskent University, Faculty of Dentistry, Department of Periodontology between January 2019 and January 2021 were reviewed. Fifty three patients were excluded due to unclear or missing data, and five subjects were not included as they were under the age of 18. The final study population therefore consisted of 142 patients (82 males/60 females).

As well as age, gender, smoking status, and frequency of tooth brushing, medical data of the patients including hypertension, hyperlipidemia, BMI, and diabetes mellitus were obtained from the patient's hospital records.

Periodontal records of the patients were obtained for six different sites (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, and disto-lingual) per tooth.

Mean ± standard deviation (SD) and median (minimum-maximum) were utilized for quantitative variables, and number of patients (percentage) were utilized for qualitative variables as descriptors. For quantitative variables, Kruskal-Wallis H test was performed to see whether there was a statistically significant difference between categories of the qualitative variable with more than two categories. Chi-square test was used for investigating the relationship between two qualitative variables. For determining the risk factors considered to have an effect on the dependent quantitative variable, univariate and multivariate logistic regression analyses were performed. Statistical significance level was defined to be 0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with periodontitis who applied to Baskent University, Faculty of Dentistry, Department of Periodontology between January 2019 and January 2021

Exclusion Criteria:

* being under the age of 18,
* being pregnant,
* having used antibiotics within the past 3 months,
* having missing data in dental and medical records.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with periodontitis who applied to Baskent University, Faculty of Dentistry, Department of Periodontology between January 2019 and January 2021
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth (PPD) | 20 minutes
  Probing pocket depth (PPD = distance between gingival margin and bottom of the periodontal pocket)were evaluated in each patient. All periodontal measurements were recorded at six sites around each tooth by a periodontal probe excluding third molar

CONTACTS AND LOCATIONS:
Overall Officials: Mehtap Bilgin Çetin, DDS,PhD, Principal Investigator — Department of Periodontology, Faculty of Dentistry, Baskent University
Locations (1):
- Baskent University,Department of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No